CLINICAL TRIAL: NCT04917393
Title: Multi-Organ Denervation to RedUce Sympathetic Drive, Multi-Center, Prospective Feasibility Study - The MODUS ON MED Study
Brief Title: Multi-Organ Denervation With the iRF System to RedUce Sympathetic Drive
Acronym: MODUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Metavention (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 2040
Record Dates: First submitted 2021-06-01; First posted 2021-06-08 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Hypertension; Type 2 Diabetes; Metabolic Syndrome
Keywords: Renal Denervation; Hepatic Denervation
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: The study is a prospective, single-arm, multi-center, sham controlled feasibility study
Who Masked: Participant
Masking Description: Subjects will be blinded during the procedure by a combination of the conscious sedation, sensory isolation and sedation and lack of familiarity of the procedural details and duration (i.e., subjects will not know the difference between the renal angiography procedure alone and the renal angiography and denervation procedure).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-organ denervation (Experimental): Multi-organ (Hepatic and Renal) denervation with the Integrated Radio Frequency (iRF) Denervation System
  Interventions: Device: iRF System Multi-organ Denervation
- Control Arm (Sham Comparator): Subjects will recieved the sham procedure
  Interventions: Other: Control Procedure

INTERVENTIONS:
Device: iRF System Multi-organ Denervation — If assigned to the treatment arm, subjects will remain blinded and recieve angiography prior to catheter based RF ablation to circumferentially disrupt the sympathetic nerves surrounding the target arteries
  Arms: Multi-organ denervation
Other: Control Procedure — If assigned to the control group, subjects will remain blinded and recieve angiography of the target arteries prior to sheath removal.
  Arms: Control Arm

SUMMARY:
The objective of the study is to evaluate the safety of multi-organ denervation using the Integrated Radio Frequency (iRF) Denervation System. and to understand any potential improvement in hypertension and glycemic control.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, multi-center, sham contollred trial to evaluate the initial safety and performance of multi-organ denervation for the treatment of hypertension and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 80 years old
2. Office systolic blood pressure (SBP) ≥ 135 mmHg or on a stable dose of antihypertensive medication(s) for at least 30 days
3. Documented daytime systolic ambulatory blood pressure (ABP) ≥ 135 and < 175 mmHg
4. HbA1c ≥7.5% - ≤11.0% on a stable dose of antidiabetic medication(s) for at least 90 days
5. Waist circumference ≥ 102 cm (male) and ≥ 88 cm (female)

   Exclusion Criteria:
6. Renal artery (RA) anatomy on either side OR common hepatic artery (CHA) anatomy, ineligible for treatment including the following:

   1. CHA OR RA artery diameter < 4.0 mm or > 7.0 mm
   2. CHA or RA length that does not allow adequate landing zone for at least one iRF balloon placement and treatment
   3. Only one functioning kidney
   4. Presence of abnormal kidney tumors
   5. CHA or RA with aneurysm
   6. Pre-existing stent or history of angioplasty in target arteries
   7. Fibromuscular dysplasia of the CHA or renal arteries
   8. Presence of CHA OR RA diameter stenosis >30%
   9. Individual lacks appropriate arterial anatomy for treatment or for maneuvering of the device from the femoral artery to the target location(s)
7. Prior renal denervation procedure
8. Type 1 diabetes mellitus
9. Use of insulin within 90 days prior to Index Procedure
10. eGFR < 45 mL/min per 1.73 m2
11. One or more documented severe hypertensive crisis (persistent or elevated hypertension > 180 mmHg accompanied by clinical symptoms) in the 90 days prior to Index Procedure
12. One or more documented hyperglycemia episodes (requiring hospitalization) in the 90 days prior to Index Procedure
13. One or more Severe hypoglycemic events (severe cognitive impairment requiring external assistance for recovery) in the 90 days prior to Index Procedure
14. Evidence of active infection within 7 days prior to Index Procedure
15. Documented history of chronic active inflammatory bowel disorders such as Crohn's disease or ulcerative colitis
16. Any history of cerebrovascular event (e.g., stroke, transient ischemic event, and cerebrovascular accident) within 6 months prior to Index Procedure
17. Myocardial infarction within 6 months of Index Procedure
18. Heart failure (New York Heart Association [NYHA] Class III-IV) at time of consent.
19. Documented confirmed episode(s) of stable or unstable angina within 6 months prior to Index Procedure
20. Documented history of persistent or permanent atrial tachyarrhythmia
21. Chronic oxygen support or mechanical ventilation other than nocturnal respiratory support for sleep apnea
22. Night shift workers
23. Chronic regular use (e.g., daily use) of NSAIDs for 6 months or greater. Aspirin therapy is allowed.
24. Active implantable medical device (e.g., ICD or CRT-D, neuromodulator/spinal stimulator, baroreflex stimulator)
25. Known Primary pulmonary hypertension (HTN) (> 60 mmHg pulmonary artery or right ventricular systolic pressure)
26. Individual has known pheochromocytoma, Cushing syndrome, primary hyperaldosteronism, coarctation of the aorta, untreated hyperthyroidism, untreated hypothyroidism, or primary hyperparathyroidism. (Note: Treated hyperthyroidism and treated hypothyroidism are permissible.)
27. A history of bariatric surgery, baroreflex activation therapy, or liver transplant, or these procedures are planned in the 365 days following Index Procedure
28. Previous hepatobiliary surgery/intervention that in the opinion of the investigator could preclude the ability to perform denervation of the CHA
29. History or diagnosis of proliferative retinopathy or advanced autonomic neuropathy (e.g., orthostatic hypotension attributable to autonomic neuropathy, a diagnosis of gastroparesis, or a clinical history strongly suggestive of delayed gastric emptying)
30. ALT or AST greater than 200 U/L
31. History or evidence of active / suspected chronic liver or biliary disease including Hepatitis B, Hepatitis C, autoimmune hepatitis, primary biliary cholangitis (PBC), primary sclerosing cholangitis, Wilson's disease, alpha-1-antitrypsin deficiency, hemochromatosis, drug-induced liver disease, bile duct dilation and obstruction, symptomatic gallstones, liver cancer or liver cirrhosis. Note: subjects with past symptomatic gallstones and a cholecystectomy are not excluded.
32. Current or chronic pancreatitis
33. Documented contraindication or allergy to contrast medium not amenable to treatment
34. Limited life expectancy of < 1 year at the discretion of the investigator
35. Any known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or for any reason in the opinion of the investigator, would be unlikely or unable to comply with study protocol requirements or whose participation may result in data analysis confounders
36. Pregnant, nursing, or planning to become pregnant (documented negative pregnancy test result required documented within a maximum of 7 days before Index Procedure for all women of childbearing potential)
37. Concurrent enrollment in any other investigational drug or device trial (participation in noninterventional registries is acceptable)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of SADEs | Index Procedure through 30 days.
  The primary safety endpoint is the incidence rate of serious adverse device effects (SADEs)

SECONDARY OUTCOMES:
Change in automated unobserved average office blood pressure | 90, 180 and 365 days
  Change from baseline in systolic/diastolic blood pressure as indicated by average automated unobserved office blood pressure
Change in Systolic/Diastolic Blood Pressure - Ambulatory Blood Pressure Monitoring | 90, 180 and 365 days
  Change from baseline in systolic/diastolic blood pressure as indicated by ambulatory blood pressure monitoring
Change in Glycemic control - HbA1c | 90 days, 180 days and 365 days
  Change from baseline in HbA1c percent
Change in Glycemic control - fasting glucose | 90 days, 180 days and 365 days
  Change from baseline in fasting plasma glucose

CONTACTS AND LOCATIONS:
Locations (2):
- Georgia (2):
  - Israeli-Georgian Medical Research Clinic Helsicore, Tbilisi
  - Tbilisi Heart and Vascular Clinic, Tbilisi

IPD SHARING:
Plan to Share IPD: Undecided